CLINICAL TRIAL: NCT01126060
Title: Efficacy of Fibrin Sealant to Reduce the Amount of Postoperative Drain in Patients With Harmonic Scalpel-assisted Total Thyroidectomy With Anterior Compartment Neck Dissections
Brief Title: Efficacy of Fibrin Sealant to Reduce the Amount of Post-thyroidectomy Drain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Man Ki Chung/Assistant professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009-12-093
Record Dates: First submitted 2010-04-15; First posted 2010-05-19 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-11

CONDITIONS: Thyroid Carcinoma; Thyroidectomy
Keywords: Neck dissection
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyroidectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Fibrin sealant (Active Comparator): usage of fibrin sealant after surgery
  Interventions: Drug: Usage of Fibrin sealant; Procedure: Thyroidectomy
- Control (No Intervention): No usage of fibrin sealant
  Interventions: Procedure: Thyroidectomy

INTERVENTIONS:
Drug: Usage of Fibrin sealant — Usage of 1 vial of fibrin sealant after hemostasis in total thyroidectomy with anterior compartment neck dissection
  Arms: Fibrin sealant
Procedure: Thyroidectomy — surgical removal of bilateral thyroid glands

SUMMARY:
Fibrin sealant has been studied to reduce post-thyroidectomy drain and hospital stay as well. However, no strong evidence from well-designed clinical trials is available. Harmonic scalpel is a ultrasonic vibrating scissors which makes it easy to cut and coagulate the tissues, thus reducing op time and postoperative drain, which is important to minimize hospital stay. The investigators hypothesized that fibrin sealant combined with harmonic scalpel-assisted procedure could guarantee no-drain postoperative care in total thyroidectomy with anterior compartment neck dissection.

ELIGIBILITY:
Inclusion Criteria:

* proven thyroid carcinoma
* Thyroidectomy with anterior compartment neck dissection

Exclusion Criteria:

* No use of harmonic scalpel during surgery
* coagulation abnormality
* refuse to participate

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2010-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Fibrin Sealant: drug used : fibrin sealant dosage : 1 vial method : spraying over surgical bed frequency : 1 vial at a time (no multiple usage)
- No Fibrin Sealant: No usage of fibrin sealant No usage of alternative drugs
Period: Overall Study
Arm/Group | Fibrin Sealant | No Fibrin Sealant
Started | 40 | 40
Completed | 40 | 38
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibrin Sealant | No Fibrin Sealant | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47.8 (9.6) | 50.8 (10.8) | 49.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 27 | 61
  Male | 6 | 13 | 19
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Drainage Amount
Description: method : measurement of drainage fluids from negative suction system every 8 hr until daily total amount reduces under 20mL
Time Frame: serial measurement from 1day to 4day after surgery
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Fibrin Sealant | No Fibrin Sealant
Number analyzed (Participants) | 38 | 40
mL | 93.5 (30.7) | 105.7 (31.2)

ADVERSE EVENTS:
Arm/Group | Fibrin Sealant | No Fibrin Sealant
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 0/38 | 0/40

LIMITATIONS AND CAVEATS:
realtive small number of patients to retrieve significant difference between two groups

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes